CLINICAL TRIAL: NCT00275119
Title: Protocole de Phase II: Etude de Faisabilite de L'Oxaliplatine en Association Chimio-Radiotherapie Concomitante Dans le Traitement Des Cancers du Pancreas Localement Avances Non Resecables
Brief Title: Gemcitabine and Oxaliplatin Followed By Radiation Therapy, Fluorouracil, and Oxaliplatin in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454568; GERCOR-D03-1; EU-20570; SANOFI-GERCOR-D03-1
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-01

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Oxaliplatin; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: oxaliplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with oxaliplatin followed by radiation therapy, fluorouracil, and oxaliplatin works in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with locally advanced, nonresectable adenocarcinoma of the pancreas treated with gemcitabine hydrochloride and oxaliplatin followed by concurrent radiotherapy, fluorouracil, and oxaliplatin.

Secondary

* Determine the tolerability of this regimen, in both the short- and long-term, in these patients.
* Determine recurrence-free survival, overall survival, and response rate in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine the clinical benefits of this regimen in these patients.
* Determine locoregional and metastatic progression-free survival of patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

* Chemotherapy: Patients receive gemcitabine hydrochloride over 100 minutes on day 1 and oxaliplatin IV over 2 hours on day 2. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are restaged at day 15-21 of the fourth course of chemotherapy. Patients with nonmetastatic disease proceed to chemoradiotherapy.
* Chemoradiotherapy: Patients undergo radiotherapy 5 days a week for 5 weeks. Patients also receive fluorouracil IV continuously in weeks 1-5 and oxaliplatin IV over 1 hour on days 1, 8, 15, 22, and 29 in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at restaging, and at day 28 after completion of chemoradiotherapy.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * Locally advanced, nonresectable disease
  * Residual disease after surgical resection (R1, R2) OR recurrent disease after radical surgery
* No visceral or peritoneal metastases
* No adenocarcinoma of the bile ducts or the ampulla of Vater

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Stable or controlled pain with analgesics
* Not pregnant or nursing
* Neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times normal OR < 3 mg/dL
* Creatinine clearance ≥ 40 mL/min
* Bilirubin ≤ 1.5 times normal
* Alkaline phosphatase < 5 times normal
* No medical condition that would preclude study treatment
* No active infection
* Negative pregnancy test
* No serious cardiac or respiratory disease
* No uncontrolled or persistent hypercalcemia
* No pre-existing neuropathy
* No biliary or gastro-duodenal obstruction
* No other malignancy except nonmelanomatous skin cancer, prostate cancer, or carcinoma in situ of the cervix or bladder
* No familial, social, geographical, or psychological condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior abdominal radiotherapy (encompassing the liver, pancreas, or spleen)
* At least 2 months since prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Tolerability
Recurrence-free survival
Overall survival
Response rate
Quality of life
Clinical benefits
Locoregional and metastatic progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Moureau-Zabotto, MD, Study Chair — Institut Paoli-Calmettes
Locations (11):
- France (11):
  - Institut Sainte Catherine, Avignon
  - Hopital Saint Andre, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Hopital Drevon, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Hopital Saint - Louis, La Rochelle
  - Clinique Victor Hugo, Le Mans
  - Clinique Saint Jean, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris

REFERENCES:
- [Result] Moureau-Zabotto L, Phelip JM, Afchain P, Mineur L, Andre T, Vendrely V, Lledo G, Dupuis O, Huguet F, Touboul E, Balosso J, Louvet C. Concomitant administration of weekly oxaliplatin, fluorouracil continuous infusion, and radiotherapy after 2 months of gemcitabine and oxaliplatin induction in patients with locally advanced pancreatic cancer: a Groupe Coordinateur Multidisciplinaire en Oncologie phase II study. J Clin Oncol. 2008 Mar 1;26(7):1080-5. doi: 10.1200/JCO.2007.12.8223. PMID 18309942
- [Result] Moureau-Zabotto L, Phélip J, Afchain P, et al.: Concomitant administration of weekly oxaliplatin, 5FU continuous infusion and radiotherapy in locally advanced pancreatic cancer (LAPC): a Gercor phase II study. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1077, S173-4, 2006.